CLINICAL TRIAL: NCT05762536
Title: A Randomized Phase II Trial of Docetaxel or Cabazitaxel With or Without Darolutamide in Men With Metastatic Castration-resistant Prostate Cancer
Brief Title: Docetaxel or Cabazitaxel With or Without Darolutamide in mCRPC
Acronym: DAROTAXEL
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Prof. R.H.J. Mathijssen, MD, PhD, Prof. dr., Erasmus Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL83539.078.23
Record Dates: First submitted 2023-02-17; First posted 2023-03-09 (Actual); Last update posted 2024-06-27 (Actual); Status verified 2024-06

CONDITIONS: Metastatic Castration-resistant Prostate Cancer
MeSH Terms: interventions — darolutamide; Docetaxel; cabazitaxel

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Docetaxel or cabazitaxel (SOC) (Active Comparator)
  Interventions: Drug: Docetaxel or cabazitaxel
- Docetaxel or cabazitaxel with darolutamide (Experimental)
  Interventions: Drug: Darolutamide; Drug: Docetaxel or cabazitaxel

INTERVENTIONS:
Drug: Darolutamide — Darolutamide 600 mg b.i.d. until the end of the last taxane cycle
  Arms: Docetaxel or cabazitaxel with darolutamide
Drug: Docetaxel or cabazitaxel — Docetaxel or cabazitaxel Q3W

SUMMARY:
Taxane efficacy in metastatic prostate cancer is modest due to resistance development. Several clinical phase III studies in metastatic castration-naïve prostate cancer (mCNPC) patients have shown that adding an androgen receptor signalling inhibitor (ARSi) to patients receiving a taxane and androgen deprivation therapy (ADT) improves survival endpoints. Adding ARSi darolutamide to docetaxel+ADT in mCNPC patients resulted in a robust OS benefit (HR 0.68). Importantly, the combination of a taxane and darolutamide is not prone to a drug-drug interaction, while there is a detrimental CYP3A4 inducing effect in the case of enzalutamide, resulting in a significant and clinically relevant reduction of cabazitaxel plasma concentrations. The investigators have previously reported preclinical data showing that addition of an androgen receptor signaling inhibitor (ARSi) improves cabazitaxel efficacy, even in metastatic castration-resistant prostate cancer (mCRPC). As treatment options for mCRPC) patients are scarce and patients often develop drug resistance relatively early, a new treatment regimen for this population to delay drug resistance is highly desired. The investigators propose a randomized phase II trial to investigate the efficacy of docetaxel or cabazitaxel plus darolutamide compared to docetaxel or cabazitaxel monotherapy in men with metastatic CRPC, who have progressed on an ARSI.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years;
2. A confirmed diagnosis of progressive mCRPC (progression according to Prostate cancer Working Group (PCWG) 3 criteria, castration defined as castrate levels of testosterone of <0.5 ng/mL) with an indication for docetaxel or cabazitaxel.
3. Patients should have had disease progression previously on at least one ARSi (abiraterone, apalutamide, darolutamide or enzalutamide). ARSi administration is allowed both in the mCNPC and in the mCRPC setting. Previous co-administration of docetaxel in mCNPC (triplet-therapy) is allowed, if patients will receive cabazitaxel in this study.
4. WHO performance ≤ 2
5. Able and willing to sign the Informed Consent Form prior to screening evaluations
6. Adequate haematological, renal and liver function and chemistry.

Exclusion Criteria:

1. Impossibility or unwillingness to take oral drugs
2. Hypersensitivity to taxanes
3. Known serious illness or medical unstable conditions that could interfere with this study requiring treatment (e.g. HIV, hepatitis, Varicella zoster or herpes zoster, organ transplants, kidney failure, serious liver disease (e.g. severe cirrhosis), cardiac and respiratory diseases)
4. Symptomatic peripheral neuropathy CTCAE grade ≥2
5. Docetaxel-rechallenge.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 245 (Estimated)
Dates: Start 2023-11-29 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first
  progression free survival, which is defined as time from randomization to radiologic, biochemical or pain progression or death from any cause, whichever occurs first, according to PCWG3

SECONDARY OUTCOMES:
Overall survival | From date of randomization until the date of death from any cause
  Overall survival, defined as time from randomization to death from any cause.
Time to progression | From date of randomization until the date of first documented progression
  Time to progression, defined as time from randomization to radiologic, biochemical or pain progression, whichever occurs first.
Time to PSA progression | From date of randomization until the date of first documented PSA progression
  Time to PSA progression, defined as time from randomization to biochemical progression.

CONTACTS AND LOCATIONS:
Locations (1):
- Erasmus MC Cancer Institute, Rotterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No